CLINICAL TRIAL: NCT06155916
Title: Sleep Structure in Neuropathic Pain Patients, Psychological Factors, Brain Connectivity, and the Effect of Pregabalin on Sleep and Pain
Brief Title: Sleep and Neuropathic Pain - Intervention Study on Pregabalin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Hanna Harno, Director, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYH2020214
Record Dates: First submitted 2023-05-29; First posted 2023-12-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Neuropathic Pain; Insomnia; Sleep Disorder
Keywords: polysomnography; actigraphy; fMRI; pregabalin; neuropathic pain
MeSH Terms: conditions — Neuralgia; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Patients start with pregabalin at dose 25mg-75mg per day according to their preference and dose will be added by 25mg to 75 mg/ 4 days up to the highest dosage the patient tolerates (maximum 300mg twice daily). After having pregabalin stabile for one month with the highest tolerated dosage, post-examinations are repeated while still using pregabalin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High ISI (Experimental): Patients that have clinically significant insomnia according to ISI questionnaire (score 15 or more) at baseline.
  Interventions: Drug: Pregabalin
- Low ISI (Experimental): Patients with no clinically significant insomnia according to ISI questionnaire (score 14 or less) at baseline.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin administration and titration to the highest dosage that the patient tolerates. The patient continues with the highest dose for one month and the pre-intervention studies are repeated.
  Other Names: Pregabalin for high insomnia patients with painful neuropathy; Pregabalin for low insomnia patients with painful neuropathy

SUMMARY:
The goal of this clinical study is to study sleep and its microstructure in neuropathic pain patients who have or who do not have a clinically significant sleep disturbance, before and during (after 1-month stabile dosage) pregabalin treatment. To find out whether reduced pain by pregabalin associates with improved sleep quality; to study, using resting state fMRI, brain network connectivity and the volume of the choroid plexus before and during pregabalin treatment (after dosage stable for one month) at baseline and during stabile treatment with pregabalin, and to compare the usability and reliability of sleep-related information collected with sleep diaries, actigraphy, iButtons, and ambulatory polysomnography in peripheral painful neuropathy patients. The main questions it aims to answer are:

* Is pregabalin more efficacious in neuropathic pain patients who suffer from insomnia compared to those with no clinically meaningful sleep disturbance?
* Does sleep disturbance due to pain associate with brain network connectivity and may these changes be reversed by pregabalin treatment? Participants will
* Fulfill e-questionnaires and keep sleep diary before and after 1month stabile pregabalin intervention
* Before and after 1-month stabile pregabalin medication: 1-week Actiwatch monitoring, iButton (1 day and night), ambulatory polysomnography (1 night), brain fMRI.

Researchers will compare patients with high ISI score patients to see if they benefit more from pregabalin treatment than those with low ISI score.

DETAILED DESCRIPTION:
This is a clinical study to analyze sleep and pain and their response to pregabalin in 40 patients aged 18 to 75 years with chronic (duration>3 months) moderate to severe pain (NRS ≥ 4/10) due to peripheral neuropathy. The investigators divide patients to two groups according to scores in ISI: the ones with clinically significant insomnia with score 15 or more (ISI High) and the ones without marked insomnia with score 14 or lower (ISI Low). Sleep will be assessed by a sleep diary, iButton, polysomnography and 1-week Actiwatch monitoring before and after 1-month stabile pregabalin dosage. Additionally, at these time points, several questionnaires regarding pain, sleep, mood, and quality of life and functional brain MRI will be performed. At pregabalin administration, the dose is added three to four day intervals, if tolerated by the patient. After a maximum tolerated dose has been stable for 1 month, the sleep studies, questionnaires, and brain fMRI are repeated. The study duration is about 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (duration > 3 months) painful peripheral neuropathy
* Pain moderate to severe (NRS ≥ 4/10) during the past week

Exclusion Criteria:

* psychotic depression, clinically significant bipolar disorder
* contraindication for performing brain fMRI (metal in the body etc)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pregabalin response to pain | Change from baseline pain intensity and interference immediately after the intervention
  Pain intensity and interference assessed by numeric rating scale
Pregabalin effect on sleep stages | Change from baseline immediately after the intervention
  1-night Ambulatory Polysomnography (NREM stage III)
Sleep disturbance associations to brain network connectivity | Change from baseline immediately after the intervention
  Brain fMRI for brain network connectivity
Sleep disturbance associations to choroid plexus volume in brain fMRI | Change from baseline immediately after the intervention
  Brain fMRI for choroid plexus volume measures
Pregabalin effect on circadian rhythms | Change from baseline immediately after the intervention
  1-week actigraphy
Pregabalin effect on body temperature during sleep | Change from baseline immediately after the intervention
  1-night body temperature measurement by iButton

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Harno, PhD, Study Chair — Helsinki University Hospital, Department of Neurology
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki, HUS
  - Helsinki University Hospital, Department of Neurology, Helsinki, Uusimaa